CLINICAL TRIAL: NCT00255619
Title: A Randomized, Multi-Center, Open Label Trial to Establish the Equivalence Between ANDY-Disc® (Fresenius Medical Care) and Ultrabag® (Baxter) in Patients on CAPD. [CAPD-2 Trial]
Brief Title: Open Label Trial to Establish the Equivalence Between ANDY-Disc® and Ultrabag® in Patients on CAPD.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ministry of Health, Malaysia (Other Government)
Collaborators: Fresenius Medical Care North America (Industry); Baxter Healthcare Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT2372
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2005-11

CONDITIONS: Chronic Renal Failure
Keywords: Continuous ambulatory peritoneal dialysis (CAPD); Peritonitis; ANDY-disc® (Fresenius Medical care); Ultra® (Baxter); Twin bag System
MeSH Terms: conditions — Kidney Failure, Chronic; Peritonitis

INTERVENTIONS:
Device: Baxter's UltraBag® and FMC Andy·Disc®

SUMMARY:
Apart from haemodialysis, continuous ambulatory peritoneal dialysis (CAPD) is another effective therapy for end stage renal disease (ESRD). The Achilles heel of CAPD however is peritonitis, which is a major cause of morbidity and mortality in CAPD patients. Advances in connectology, such as the disconnect system, have resulted in reduced rate of peritonitis. The disconnect system which incorporated a Y-connection allow contamination occurring at the time of connection of the system to flush into the drainage bag thereby reducing the size of microorganism innoculum entering the peritoneal cavity. In recent years, the twin bag system where both the infusion and drainage bags are pre-attached to the Y tubing, has resulted in further reduction in peritonitis rate.

Two different twin bags systems are being introduced into the MOH hospitals. They are Baxter UltraBag® and Fresenius Andy·Disc®.

Even though both the systems are very similar, our own experience suggest that minor variation in the connectology could translate into marked differences in the peritonitis rate. In this multi centre, randomised controlled study, both the twin bag systems will be evaluated to establish their equivalence with respect to the incidence of peritonitis and technique failure.

DETAILED DESCRIPTION:
This is a multi-centre, open label, parallel group randomized trial designed to demonstrate the therapeutic equivalence of ANDY-Disc® with Ultrabag® for a treatment period of 12 months. 270 patients on CAPD from 6 participating sites who met inclusion/exclusion criteria were enrolled into the trial. After initial screening, patients attended clinic for baseline examination, including clearance studies. Subjects were then randomly allocated to ANDY-Disc® or Ultrabag® in a ratio of 1:1. Study visits occurred every 2 weeks through 4 weeks, then every 4 weeks through 12 weeks, and every 12 weeks thereafter for the duration of the study (12 months). Hence there were a total of 7 visits (1 screen/baseline, 2 biweekly, 2-4 weekly and 2-6 monthly treatment visits, the last being the final visit).

Safety and tolerability assessments consisted of monitoring adverse events and serious adverse events, monitoring of haematology, blood chemistry and regular performance of physical examinations.

Criteria for evaluation:

Efficacy: Primary efficacy parameter:The primary efficacy variable will be the incidence of peritonitis. Peritonitis is defined as the presence of at least two of the following

1. Abdominal pain or tenderness
2. Presence of white blood cells in peritoneal effluent in excess of 100 cells per mL composed of at least 50% polymorphs
3. Positive cultureSecondary efficacy parameter:

The secondary efficacy variables are:

1. Technique failure; defined as transfer to haemodialysis or death. Note that cross-over to a comparator treatment will be considered as withdrawal.

Frequency of technical problem or product defect, satisfaction with and difficulty in using the connection system. Technical problem and product defect shall be observed and evaluated by patient and data recorded by using a patient's diary. Satisfaction with and difficulty in using the connection systems will be evaluated by investigator in global fashion through a questionnaire.

Safety: Safety and tolerability assessments will consist of

1. Monitoring and recording all adverse events and serious adverse events.
2. Regular performance of physical examinations, including vital signs.
3. Regular monitoring of haematology and blood chemistry parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from patient or parents/guardian.
2. New or existing patients (on the single bag system) with end stage renal failure in the MOH CAPD programme with indications for using the twin bag system. For the purpose of this trial, these indications are:

   * All paediatric patients (up to the age of 18 years)
   * Patients who could not be trained to use the single bag system
   * Existing CAPD patients on the single bag system with recurrent peritonitis
   * Existing CAPD patients on the single bag system who for various reasons could no longer continue with the system.
   * Existing CAPD patients on the single bag system who in the opinion of the investigator would benefit from a switch to the twin bag system.

Exclusion Criteria:

1. Participation in any CAPD trial in which the patient received an investigational product within 30 days preceding the screening phase of this study.
2. Those persons directly involved in the conduct of the study.
3. History of non-compliance to medical regimen or patients who are unwilling or unable to comply with the protocol.
4. Any serious medical conditions or disability, which in the opinion of the investigator, would interfere with treatment or assessment or preclude completion of this study.
5. Patients expected to be transferred to a non participating centre within the next six months
6. Patients presently on a twin bag system
7. Use of automated cycler assistance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 264
Dates: Start 2002-05; Study Completion 2004-05

PRIMARY OUTCOMES:
To establish the equivalence of ANDY-disc® with Ultrabag® for a treatment period of 12 months in patients on CAPD with respect to peritonitis rate.

SECONDARY OUTCOMES:
To compare ANDY-disc® with Ultrabag® with respect to technique failure
To compare ANDY-disc® with Ultrabag® with respect to their respective frequency of technical problem or product defect, satisfaction with and difficulty in using the connection system.

CONTACTS AND LOCATIONS:
Overall Officials: Zaki Morad, MRCP, FRCP, Principal Investigator — Ministry of Health
Locations (6):
- Malaysia (6):
  - Department of Medicine, Sultanah Aminah Hospital, Johor Bharu, Johor
  - Department of Nephrology, Kuala Lumpur Hospital, Kuala Lumpur, Kuala Lumpur
  - Department of Pediatrics, Kuala Lumpur Hospital, Kuala Lumpur, Kuala Lumpur
  - Department of Medicine, Seremban Hospital, Seremban, Negeri Sembilan
  - Department of Medicine, Penang Hospital, George Town, Pulau Pinang
  - Department of Nephrology,Selayang Hospital, Selayang Baru Utara, Selangor

REFERENCES:
- See also: the link is an academic research organisation for the trial — http://www.crc.gov.my